CLINICAL TRIAL: NCT01477970
Title: Double GnRH Antagonist Daily Dose in Hyperresponding IVF/ICSI Cycles May Prevent the OHSS
Status: Completed | Type: Observational
Sponsor: Iakentro Fertility Centre (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Yannis Prapas, Associated Professor, Iakentro Fertility Centre
Other Study IDs: abcd1234
Record Dates: First submitted 2011-06-30; First posted 2011-11-23 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: GnRH antagonists; OHSS; ovarian stimulation
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The possibility to prevent the early ovarian hyperstimulation syndrome (OHSS) by doubling the daily dose of GnRH-antagonist in women stimulated with the antagonist protocol who are at risk for OHSS was evaluated. Thirty-eight women of a study group who underwent ovarian stimulation using the GnRH-antagonist protocol and might have had their cycle cancelled because of OHSS were compared to 76 women of a control group. All cases of the study group were IVF women presenting a rapid rise of E2 ≥ 3500 pg/ml on the 7th day of stimulation or later while the follicles (> 12mm) were > 15 in total and the biggest one was ≤ 16mm in diameter. By decreasing the rFSH dose to 100IU a day and adding an additional dose of GnRH-antagonist (0.25 twice a day), estradiol levels were lowered or reached a plateau before hCG was given. A marked decrease or plateau of estradiol levels was observed the day of oocyte retrieval while the pregnancy rate was not adversely affected when compared with an optimum ovarian response cycles. None of the women were cancelled or developed OHSS.

In overresponding IVF cycles, doubling the usual GnRH-antagonist daily-dose during the ovarian stimulation, the estradiol rise could be blocked while a minimal follicular stimulation may continue without the risk of OHSS or adversely affect pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Women stimulated with the antagonist protocol who are at risk of ovarian hyperstimulation syndrome

Exclusion Criteria:

* Has chosen other preventive protocols (coasting and/or cryopreservation)were excluded

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: PILOT STUDY
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)